CLINICAL TRIAL: NCT02096081
Title: The Treatment of Glabellar Frown Lines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUS 60201_4096_1
Record Dates: First submitted 2014-03-20; First posted 2014-03-26 (Estimated); Results first posted 2017-03-16 (Actual); Last update posted 2017-10-19 (Actual); Status verified 2017-09

CONDITIONS: Glabellar Frown Lines
Keywords: Glabellar Frown Lines; Frown Lines; Facial Wrinkles
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IncobotulinumtoxinA (Experimental): 20U injection: equal aliquots of 0.1 mL (4U) to 5 injection points
  Interventions: Drug: IncobotulinumtoxinA
- OnabotulinumtoxinA (Active Comparator): 20U injection: equal aliquots of 0.1 mL (4U) to 5 injection points
  Interventions: Drug: OnabotulinumtoxinA

INTERVENTIONS:
Drug: IncobotulinumtoxinA — 20U injection: equal aliquots of 0.1 mL (4U) to 5 injection points; mode of application: intramuscular injection
  Other Names: Xeomin®; NT201; Botulinum toxin type A [150 kDa], free from complexing proteins
  Arms: IncobotulinumtoxinA
Drug: OnabotulinumtoxinA — 20U injection: equal aliquots of 0.1 mL (4U) to 5 injection points; mode of application: intramuscular injection
  Other Names: Botox®
  Arms: OnabotulinumtoxinA

SUMMARY:
The purpose of this study is to show that two FDA-approved botulinum toxin drugs called Xeomin® and Botox® can reduce the severity of vertical lines (wrinkles) that appear between the eyebrows (glabellar frown lines).

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, parallel group clinical study to investigate the equivalence of incobotulinumtoxinA (Xeomin®) to onabotulinumtoxinA (Botox®) in the treatment of glabellar frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient females 18 to 50 years of age
* Moderate to severe glabellar frown lines

Exclusion Criteria:

* Glabellar Frown Lines at rest rating 3 on the 4-point Facial Wrinkle Scale
* Previous treatment with botulinum toxin
* Previous treatment with biodegradable fillers in glabellar area within last 12 months
* Any severe or uncontrolled systemic disease, malignant tumor, or medical history of HIV infection
* Known hypersensitivity to incobotulinumtoxinA or onabotulinumtoxinA or to any of their excipients
* Intake of any of the forbidden concomitant medication or other agents that might interfere with neuromuscular function or might interfere with the action of botulinum toxin type within 14 days prior to injection

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Schlӧbe, MD, Study Director — Merz North America, Inc.
Locations (10):
- United States (10):
  - Merz Investigative Site #001099, Los Angeles, California
  - Merz Investigative Site #001300, Sacramento, California
  - Merz Investigative Site #001299, Santa Monica, California
  - Merz Investigative Site #001298, Washington D.C., District of Columbia
  - Merz Investigative Site #001170, Washington D.C., District of Columbia
  - Merz Investigative Site #001101, Coral Gables, Florida
  - Merz Investigative Site #001105, Metairie, Louisiana
  - Merz Investigative Site #001098, Chestnut Hill, Massachusetts
  - Merz Investigative Site #001297, New York, New York
  - Merz Investigative Site #001097, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kane MA, Gold MH, Coleman WP 3rd, Jones DH, Tanghetti EA, Alster TS, Rohrer TE, Burgess CM, Shamban AT, Finn E. A Randomized, Double-Blind Trial to Investigate the Equivalence of IncobotulinumtoxinA and OnabotulinumtoxinA for Glabellar Frown Lines. Dermatol Surg. 2015 Nov;41(11):1310-9. doi: 10.1097/DSS.0000000000000531. PMID 26509943

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Started | 122 | 128
Completed | 119 | 124
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) was used and is defined as the subset of all enrolled subjects who receive the study medication. Subjects in the SES were summarized according to the treatment they received and not by the treatment to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA | Total
Number analyzed (Participants) | 122 | 128 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.3 (7.4) | 39.4 (7.8) | 39.3 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 128 | 250
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 35 | 58
  Not Hispanic or Latino | 99 | 93 | 192
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 13 | 27
  White | 104 | 107 | 211
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Measured as the Percentage of Participants Who Responded to Treatment
Description: Response defined as ≥ 1 point improvement from baseline (prior to treatment) on the Facial Wrinkle Scale at maximum frown as rated by an independent masked panel of physicians specifically qualified to assess study photographs using subject photographs at 1 month from treatment.
Time Frame: 1 Month from baseline
Population: All efficacy analyses were performed on the per protocol set (PPS) defined as the subset of subjects in the FAS for whom no major protocol deviations were identified.
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 95.7 | 99.2
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; With assumptions of an alpha of 5%, an equivalence margin of 15% for each side, the real response rate expected as 90% for incobotulinumtoxinA and onabotulinumtoxinA at day 30 and a 1:1 allocation ratio, a total of 225 subjects were needed to achieve a statistical power of 90% in order to make an equivalence conclusion at day 30. Results are based on the Newcombe-Wilson confidence interval. To account for exclusions from the PPS of about 10%, approximately 250 subjects were enrolled; Test type: Non-Inferiority or Equivalence — The analysis of response defined as the difference (D) in response rates between two treatment groups at 1 month was as follows: D = response rate in the incobotulinumtoxinA group minus the response rate in the onabotulinumtoxinA group. The hypothesis testing procedure to test the equivalence of the two products is as follows: Ho (null): D ≤ -∆ OR D ≥ ∆ versus Ha (alternate): -∆ < D < ∆, where ∆ is the margin of equivalence = 0.15; Difference in proportions of response = -3.5, 95% CI 2-sided [-7.5 to 0.6] — If the confidence interval lies within the limits of ±0.15, then Ho is rejected in favor of Ha (i.e., equivalence of incobotulinumtoxinA and onabotulinumtoxinA can be concluded); otherwise, treatment equivalence cannot be concluded

2. Secondary Outcome: Response at Maximum Frown Rated by Independent Rater
Description: Response defined as ≥ 1 point improvement from baseline on the Facial Wrinkle Scale (0=None to 3=severe) at maximum frown as rated by an independent masked panel of physicians specifically qualified to assess study photographs using subject photographs at 2 months from baseline.
Time Frame: 2 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 89.7 | 95.0
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; The study was not powered for this secondary endpoint; Test type: Non-Inferiority or Equivalence — This secondary analysis was performed for exploratory purposes. The analysis of response defined as the difference (D) in response rates between two treatment groups at 2 months was as follows: D = response rate in the incobotulinumtoxinA group minus the response rate in the onabotulinumtoxinA group; Difference in proportion of responders = -5.3, 95% CI 2-sided [-12.1 to 1.5] — If the confidence interval lies within the limits of ±0.15, then both incobotulinumtoxinA and onabotulinumtoxinA have similar efficacy profiles

3. Secondary Outcome: Response at Maximum Frown Rated by Independent Rater
Description: Response defined as ≥ 1 point improvement from baseline on the Facial Wrinkle Scale (0=None to 3=severe) at maximum frown as rated by an independent masked panel of physicians specifically qualified to assess study photographs using subject photographs at 3 months from baseline.
Time Frame: 3 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 80.2 | 80.7
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; The study was not powered for this secondary endpoint; Test type: Non-Inferiority or Equivalence — This secondary analysis was performed for exploratory purposes. The analysis of response defined as the difference (D) in response rates between two treatment groups at 3 months was as follows: D = response rate in the incobotulinumtoxinA group minus the response rate in the onabotulinumtoxinA group; Difference in proportion of responders = -0.5, 95% CI 2-sided [-10.6 to 9.6] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Response at Maximum Frown Rated by Independent Rater
Description: Response defined as ≥ 1 point improvement from baseline on the Facial Wrinkle Scale (0=None to 3=severe) at maximum frown as rated by an independent masked panel of physicians specifically qualified to assess study photographs using subject photographs at 4 months from baseline.
Time Frame: 4 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 62.1 | 67.2
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; The study was not powered for this secondary endpoint; Test type: Non-Inferiority or Equivalence — This secondary analysis was performed for exploratory purposes. The analysis of response defined as the difference (D) in response rates between two treatment groups at 4 months was as follows: D = response rate in the incobotulinumtoxinA group minus the response rate in the onabotulinumtoxinA group; Difference in proportion of responders = -5.2, 95% CI 2-sided [-17.4 to 7.1] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Response at Maximum Frown Rated by Treating Physician
Description: Response defined as ≥ 1 point improvement from baseline on the Facial Wrinkle Scale (0=None to 3=severe) at maximum frown as rated by the treating physicians using subject photographs at 1 month from treatment.
Time Frame: 1 month from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 93.1 | 95.8
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; The study was not powered for this secondary endpoint; Test type: Non-Inferiority or Equivalence — This secondary analysis was performed for exploratory purposes. The analysis of response defined as the difference (D) in response rates between two treatment groups at 1 month was as follows: D = response rate in the incobotulinumtoxinA group minus the response rate in the onabotulinumtoxinA group; Difference in proportion of responders = -2.7, 95% CI 2-sided [-8.5 to 3.2] — [estimate comment as in outcome 2, analysis 1]

6. Secondary Outcome: Response at Maximum Frown Rated by Treating Physician
Description: Response defined as ≥ 1 point improvement from baseline on the Facial Wrinkle Scale (0=None to 3=severe) at maximum frown as rated by the treating physicians using subject photographs at 2 months from treatment.
Time Frame: 2 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 87.1 | 89.9
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; The study was not powered for this secondary endpoint; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Difference in proportion of responders = -2.8, 95% CI 2-sided [-11.0 to 5.3] — [estimate comment as in outcome 2, analysis 1]

7. Secondary Outcome: Response at Maximum Frown Rated by Treating Physician
Description: Response defined as ≥ 1 point improvement from baseline on the Facial Wrinkle Scale (0=None to 3=severe) at maximum frown as rated by the treating physicians using subject photographs at 3 months from treatment.
Time Frame: 3 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 75.0 | 76.5
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; The study was not powered for this secondary endpoint; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Difference in proportion of responders = -1.5, 95% CI 2-sided [-12.4 to 9.5] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Response at Maximum Frown Rated by Treating Physician
Description: Response defined as ≥ 1 point improvement from baseline on the Facial Wrinkle Scale (0=None to 3=severe) at maximum frown as rated by the treating physicians using subject photographs at 4 months from treatment.
Time Frame: 4 months from baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
percentage of participants | 58.6 | 60.5
Statistical Analysis 1: Comparison: IncobotulinumtoxinA vs OnabotulinumtoxinA; The study was not powered for this secondary endpoint; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 4, analysis 1]; Difference in proportion of responders = -1.9, 95% CI 2-sided [-14.4 to 10.7] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Subject Satisfaction
Description: Assessment of subject treatment satisfaction by subject questionnaire and diary at 1 month from treatment. Extremely satisfied, satisfied, and slightly satisfied were categorized as "Satisfaction" and extremely dissatisfied, dissatisfied, and slightly dissatisfied were categorized as "Dissatisfaction." Subjects with missing data were categorized as "Missing."
Time Frame: 1 month from baseline
Population: This endpoint was analyzed using observed cases in the per protocol set (PPS), defined as the subset of subjects in the FAS from whom no major protocol deviations were identified.
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
participants
  Satisfaction | 112 | 116
  Dissatifaction | 3 | 3
  Missing | 1 | 0

10. Secondary Outcome: Subject Satisfaction
Description: Assessment of subject treatment satisfaction by subject questionnaire and diary at 2 months from treatment. Extremely satisfied, satisfied, and slightly satisfied were categorized as "Satisfaction" and extremely dissatisfied, dissatisfied, and slightly dissatisfied were categorized as "Dissatisfaction." Subjects with missing data were categorized as "Missing."
Time Frame: 2 months from baseline
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
participants
  Satisfied | 110 | 113
  Dissatisfied | 5 | 6
  Missing | 1 | 0

11. Secondary Outcome: Subject Satisfaction
Description: Assessment of subject treatment satisfaction by subject questionnaire and diary at 3 months from treatment. Extremely satisfied, satisfied, and slightly satisfied were categorized as "Satisfaction" and extremely dissatisfied, dissatisfied, and slightly dissatisfied were categorized as "Dissatisfaction." Subjects with missing data were categorized as "Missing."
Time Frame: 3 months from baseline
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
participants
  Satisfaction | 108 | 108
  Dissatisfaction | 7 | 10
  Missing | 1 | 1

12. Secondary Outcome: Subject Satisfaction
Description: Assessment of subject treatment satisfaction by subject questionnaire and diary at 4 months from treatment. Extremely satisfied, satisfied, and slightly satisfied were categorized as "Satisfaction" and extremely dissatisfied, dissatisfied, and slightly dissatisfied were categorized as "Dissatisfaction." Subjects with missing data were categorized as "Missing."
Time Frame: 4 months from baseline
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
participants
  Satisfaction | 107 | 104
  Dissatisfaction | 8 | 11
  Missing | 1 | 4

13. Secondary Outcome: Subject Perception of Treatment Onset
Description: Assessment of subject perception of date of treatment onset using a take-home diary
Time Frame: Open-ended time frame for the 4 month study duration. Data for onset and peak effect is recorded in the subject diary.
Population: as for outcome 9
Measure: Median (Full Range); unit: days
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
days | 3.0 [1 to 14] | 3.0 [1 to 14]

14. Secondary Outcome: Subject Perception of Treatment Peak Effect
Description: Assessment of subject perception of date of treatment peak effect using a take-home diary
Time Frame: Open-ended time frame for the 4 month study duration. Data for onset and peak effect is recorded in the subject diary.
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Number analyzed (Participants) | 116 | 119
participants
  Within 4 weeks | 108 | 113
  Longer than 4 weeks | 7 | 4
  Missing | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the entire study period (4 months). Adverse events were not followed-up after the final study visit/safety visit, which was scheduled for 4 months post-treatment.
Groups:
- IncobotulinumtoxinA: 20U injection: equal aliquots of 0.1 mL (4U) to 5 injection points.
  IncobotulinumtoxinA: 20U/injection: equal aliquots of 0.1 mL (4U) to 5 injection points; mode of application: intramuscular injection
- OnabotulinumtoxinA: 20U injection: equal aliquots of 0.1 mL (4U) to 5 injection points.
  OnabotulinumtoxinA: 20U/injection: equal aliquots of 0.1 mL (4U) to 5 injection points; mode of application: intramuscular injection
Arm/Group | IncobotulinumtoxinA | OnabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 1/122 | 1/128
Other Adverse Events (participants affected / at risk) | 9/122 | 8/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IncobotulinumtoxinA (N=122) | OnabotulinumtoxinA (N=128)
Human ehrlichiosis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IncobotulinumtoxinA (N=122) | OnabotulinumtoxinA (N=128)
Headache (Nervous system disorders) | 7 (7) | 5 (5)
Facial Asymmetry (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No